CLINICAL TRIAL: NCT06578273
Title: Peripheral Sensory Stimulation of the Hand and Synchronized Deep Breathing in the Treatment of Parkinson's Disease: Assessing Safety and Feasibility
Brief Title: NeuroGlove PD Study Clinical
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NeuroGlove LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: REG-1010
Record Dates: First submitted 2024-08-23; First posted 2024-08-29 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a prospective, homebased, interventional clinical study in which 8 subjects will be enrolled. Eight (8) subjects who suffer from Parkinson's disease will receive treatment using the NeuroGlove.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- single arm (Experimental): Subjects in the study will use NeuroGlove 60 minutes twice per day, 30 minutes to each hand. Subjects will be instructed on coordinating their breathing with device on/off periods to maximize relaxation. Subjects who complete less than 45 minutes of treatment per day will be considered noncompliant and may be replaced.
  Interventions: Device: NeuroGlove

INTERVENTIONS:
Device: NeuroGlove — The NeuroGlove is a plastic chamber with multiple apertures along its length to allow for puffs of air to be directed to the volar surface of the distal forearm, the palm, and the fingers. The NeuroGlove is intended to provide peripheral sensory stimulation to the hand through pneumatic puffs of air to encourage collateral blood supply and sensorimotor development. A pneumatic pump delivers intermittent puffs of air cycling between one second on and two seconds off. The hand with the palm facing up is placed within the device chamber on a gel pad to provide a comfortable resting surface for the duration of the treatment, which lasts approximately thirty minutes.
  The device facilitates the rehabilitation, improvement, or restoration of motion in patients with neurological disorders.

SUMMARY:
Safety and Feasibility of Peripheral Sensory Stimulation of the Hand in the Treatment of Parkinson's Disease

DETAILED DESCRIPTION:
This is a prospective, homebased, interventional clinical study in which 8 subjects will be enrolled. Eight (8) subjects who suffer from Parkinson's disease will receive treatment using the NeuroGlove.

Up to 8 subjects enrolled and complete study procedures. There will be a single cohort in the study consisting of the subjects with PD who will receive treatment with NeuroGlove.

ELIGIBILITY:
Inclusion Criteria:

1. Able to and willing to provide informed consent. Legally authorized representatives (LARs) will not be allowed to consent on behalf of the subject.
2. Men and women ≥18 and <85 years of age.
3. Carry an active diagnosis of PD
4. Suffer from PD symptoms that impact subject's daily activities and quality of life

   Exclusion Criteria:
5. Physical limitations of the upper extremity (e.g., fracture, joint deformity, severe spasticity/contracture, wounds, skin breakdown, lymphedema, etc.)
6. Lacks the ability to comprehend or follow instructions, or for any reason, in the opinion of the investigator, would be unlikely or unable to comply with study protocol requirements.
7. Currently participating in another interventional clinical trial (observational clinical trial participation is allowed for study enrollment.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-08-22 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Use the UPDRS to Evaluate safety and feasibility of device | 4 weeks
  Evaluate safety and feasibility of device use on subjects with active symptoms, monitoring motor symptoms and subjects' sense of well-being. The UPDRS - United Parkinson's Disease Rating scale - developed for research and clinical evaluation will be used. The form has a severity scale with ratings from 0-4 with 0 meaning no severity and 4 meaning extreem severity
Use Custom Satisfaction Scale to Rate and severity of adverse events related to the use of the NeuroGlove. | 4 weeks
  The Satisfaction scale will assess ease of use, satisfaction, feelings of symptom reduction among other questions with a 5 point scale: Strongly Agree, Agree, Neutral, Disagree, and Strongly Disagree

CONTACTS AND LOCATIONS:
Locations (1):
- NeuroGlove, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided